CLINICAL TRIAL: NCT04707612
Title: VDR SNPs & 25OHD Correlated With Dyslipidemia
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Chronic Disease Control (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Ji-Chang, Director of Molecular Biology Laboratory, Shenzhen Center for Chronic Disease Control
Other Study IDs: QLS2015
Record Dates: First submitted 2021-01-10; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Dyslipidemias; Single Nucleotide Polymorphism
Keywords: gene polymorphism; vitamin D receptor; vitamin D; lipid; dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples were collected for plasma or serum and DNA isolations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
The project was aimed to explore the associations of single nucleotide polymorphisms (SNPs) of vitamin D receptor gene with specific circulating lipids in adult Chinese. The circulating 25-hydroxyvitamin D concentration was also tested to explore its interactions with SNPs in the associations.

ELIGIBILITY:
Inclusion Criteria:

* 1) ≥ 20 years old Han Chinese;
* 2) living in Shenzhen for > 2 years;
* 3) free of liver diseases, renal diseases, and any cancers in the past 6 months; and
* 4) not in pregnancy for women.

Exclusion Criteria:

* 1) had severe organic diseases,
* 2) had acute infection symptoms, allergic diseases, and malignant tumors,
* 3) had a family history of genetic diseases,
* 4) took VD supplements in the past 6 months,
* 5) took medicines to control lipid levels within 12 hours, or
* 6) took diuretics, did strenuous exercise, or overate within 24 hours before the test.

Ages: 20 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers visiting a health examination center in Shenzhen city of Guangdong province, China were recruited.
  A total of 1,987 adults were included in the analysis, aged from 20 to 81 years old. Among them, there were 1,124 females aged 39 (31 - 49) years old and 863 males aged 36 (30 - 44) years old.
Sampling Method: Probability Sample
Enrollment: 1987 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
SNPs of VDR | 6 months
  Polymorphisms of vitamin D receptor gene: Cdx2, Fok1, Apa1, and Taq1
lipid profiles | 6 months
  Serum concentrations of TG, TC, LDLC, and HDLC
25OHD | 6 months
  Plasma 25-hydroxyvitamin D concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Center for Chronic Disease Control, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided